CLINICAL TRIAL: NCT02331355
Title: VCA (Hand Transplantation): Functional and Quality of Life Outcomes
Brief Title: Hand Transplantation: Functional and Quality of Life Outcomes
Status: Withdrawn | Type: Observational
Why Stopped: unable to find appropriate candidates
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Kagan Ozer, Associate Professor, University of Michigan
Other Study IDs: HUM00078607
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Amputation; Traumatic, Arm, Upper, Between Shoulder and Elbow; Amputation; Traumatic, Hand; Amputation; Traumatic, Hand, Both; Amputation; Traumatic, Arm: Forearm, at Elbow Level; Amputation; Traumatic, Arm, Upper
Keywords: amputation, hand, forearm, arm, traumatic, transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is an urgent need to develop hand transplant programs in this country. To this end, the University of Michigan Hospital and Health Systems is developing such an interdisciplinary program. The Transplant Center would like to track the patient experience from pre-operative care through surgery and post-operative care.

Detailed information will be collected from the patient medical records, including: Pre-operative screening, demographics, medications; Surgical information ; Post-operative inpatient and out-patient care; laboratory and other test results; physical assessments, psychological assessments and quality of life assessments.

DETAILED DESCRIPTION:
Vascularized composite tissue allotransplantation (VCA) is the transplantation of multiple tissues containing skin, muscle, bone, joint, cartilage, nerve, tendon, vessels. VCA is useful for functional restoration of patients with severe tissue loss as encountered with massive burns, traumatic injuries, congenital anomalies, and following tumor resection. VCA, and specifically hand transplantation, combines the technical excellence of hand surgery/microsurgery with the complex multidisciplinary care rendered in modern solid organ transplantation. The technical demands of hand transplantation, enhanced donor antigen burden of the hand allograft, and complex psychosocial issues pertaining to the recipient account for much of the discrepancy between these 2 related fields.

Detailed information will be collected from the patient medical records, including: Pre-operative screening, demographics, medications; surgical information ; post-operative inpatient and out-patient care; laboratory and other test results; physical assessments, psychological assessments and quality of life assessments.

Specific outcomes will include allograft survival, allograft rejection, allograft functionality, and quality of life from transplant through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been evaluated and listed for hand transplantation will be approached to participate in this study.

Exclusion Criteria:

* Those deemed not to be appropriate for listing by the University of Michigan interdisciplinary evaluation team.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had traumatic hand transplantation below the elbow.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Allograft survival | Transplant through end of study (5 years)
  Graft survival will be evaluated at transplant, days 14, then monthly in year 1, then yearly years 2-5

SECONDARY OUTCOMES:
Immunosuppression requirements | Transplant through end of study (5 years)
  immunosuppression will be documented throughout study
Allograft rejection | Transplant through end of study (5 years)
  Skin and muscle biopsies will be performed days 14, then monthly in year 1, then yearly years 2-5. Donor specific antibody will also be measured at these timepoints
Allograft Function | Transplant through end of study (5 years)
  Outcomes questionnaires will be completed by patient at post-transplant 3, 6, 12 months, and every year thereafter up to 5 years
Quality of life | Transplant through end of study (5 years)
  SF-36 survey results will be collected before transplant and at various time points post transplant

OTHER OUTCOMES:
Cost and utilization information | Transplant through end of study (5 years)
  cost and utilization of service will be tracked

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States